CLINICAL TRIAL: NCT03837223
Title: RESCUE PROTOCOL AND FRESH EMBRYO TRANSFER AFTER TRIGGER WITH ANALOGS OF GNRH: THE HUMANITAS PROTOCOL
Brief Title: RESCUE PROTOCOL AND FRESH EMBRYO TRANSFER
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: trigger
Record Dates: First submitted 2019-02-08; First posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: GnRH Trigger and Rescue Protocol
MeSH Terms: interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients underwent "rescue protocols" and fresh embryotransfer: they were patients with good prognosis with a mean age of 34.13 ± 4.42 years, with a good ovarian reserve
  Interventions: Drug: GnRH agonist

INTERVENTIONS:
Drug: GnRH agonist — In High Responder patients (HR) (more than 18 follicles with diameter ≥ 12mm at ovulation induction), the trigger was obtained with triptorelin 0.2 mg sc. In this cohort if less of 18 oocytes were retrieved, patients were considered at intermediate risk of OHSS and fresh transfer was performed. An adequate support of the luteal phase was initiated: HCG 1500 IU / sc the day of the pick up + estradiol 4 mg + vaginal progesterone 400 mg daily (Rescue protocol).
  Other Names: GnRH trigger

SUMMARY:
Ovarian Hyperstimulation Syndrome (OHSS) is one of the most dangerous complications of Assisted Reproductive Technologies (ART) cycles. The use in clinical practice of the GnRH antagonist has made it possible to perform the trigger with GnRH analogues reducing the risk of OHSS. The trigger with analogue increases the Abortion Rate (AR) and reduces the Ongoing Pregnancy Rate (OPR), because the luteal phase in these cycles is particularly deficient. To reduce this occurrence several studies have focused on the importance of support of the luteal phase. The aims of study is to evaluate OPR and AR in patients at intermediate risk of OHSS (<18 recovered oocytes) which performed GnRH trigger and rescue protocol.

ELIGIBILITY:
Inclusion Criteria:

AMH ( antimullerian hormone) > 3.5 ng / ml, AFC (antral follicles count) > 15 follicles and if more than 18 follicles with diam. 12mm to induction

Exclusion Criteria:

high risk of OHSS ( ovarian hyperstimulation syndrome)

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: In HR patients (AMH> 3.5 ng / ml, AFC> 15 follicles and if more than 18 follicles with diam. 12mm to induction) the trigger was obtained with triptorelin 0.2 mg / sc. In patients considered to be at intermediate risk of OHSS a rescue protocol has been implemented (HCG 1500 IU / sc the day of the pick up + estradiol 4 mg + vaginal progesterone 400 mg daily) and fresh embryo transfer.
Sampling Method: Non-Probability Sample
Enrollment: 271 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
ongoing pregnancy rate (OPR) | 2013-2018
  presence of gestational sac and fetal hearts beats showed on unltrasonography 7/8 weeks after embryo transfer

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kupka MS, Ferraretti AP, de Mouzon J, Erb K, D'Hooghe T, Castilla JA, Calhaz-Jorge C, De Geyter C, Goossens V; European IVF-Monitoring Consortium, for the European Society of Human Reproduction and Embryology. Assisted reproductive technology in Europe, 2010: results generated from European registers by ESHREdagger. Hum Reprod. 2014 Oct 10;29(10):2099-113. doi: 10.1093/humrep/deu175. Epub 2014 Jul 27. PMID 25069504
- [Result] Humaidan P, Kol S, Papanikolaou EG; Copenhagen GnRH Agonist Triggering Workshop Group. GnRH agonist for triggering of final oocyte maturation: time for a change of practice? Hum Reprod Update. 2011 Jul-Aug;17(4):510-24. doi: 10.1093/humupd/dmr008. Epub 2011 Mar 30. PMID 21450755
- [Result] Fatemi HM, Garcia-Velasco J. Avoiding ovarian hyperstimulation syndrome with the use of gonadotropin-releasing hormone agonist trigger. Fertil Steril. 2015 Apr;103(4):870-3. doi: 10.1016/j.fertnstert.2015.02.004. Epub 2015 Feb 24. PMID 25724740